CLINICAL TRIAL: NCT02302690
Title: Study of the Prevalence of Pre-existing Immunity Against the Adeno-associated Virus (AAV) in Patients With Crigler-Najjar Syndrome
Brief Title: Immunity Against AAV in Crigler Najjar Patient
Status: Completed | Type: Observational
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Other Study IDs: CRIG-COL-01
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Crigler Najjar Syndrome
MeSH Terms: conditions — Crigler-Najjar Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Blood sample for immunology

SUMMARY:
The proposed research protocol aims at addressing these points by pre-screening CN patients for their AAV serology in link with their medical history and current medical status. A first objective is to assess the presence of neutralizing AAV antibodies in the serum of CN patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a Crigler-Najjar syndrome
* The molecular diagnosis has been confirmed by UGT1A1 gene DNA sequencing

Exclusion criteria:

* The patient is liver transplanted
* The patient is suffering from severe associated pathologies precluding further enrolment in a future interventional clinical study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Crigler Najjar syndrome
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To assess the presence of neutralizing AAV antibodies in the serum of CN patients | 1 day visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Antoine Béclère, Clamart, France